CLINICAL TRIAL: NCT03020329
Title: Phase II Study of TPF Induction Chemotherapy Followed by Concurrent Chemoradiotherapy in Young Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy in Young Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor and Deputy Director, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC in Young Patients
Record Dates: First submitted 2016-12-14; First posted 2017-01-13 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Nasopharyngeal Carcinoma; Children
Keywords: Induction Chemotherapy; Nasopharyngeal carcinoma; Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Drug Therapy; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel liposome, Cisplatin, 5-Fu, (Experimental): Patients receive paclitaxel liposome(135mg/m2 on day 1), cisplatin (75mg/m2 on day 1,Separate injection on day 1 to 3) and fluorouracil (3750mg/m2 CIV 120h) every three weeks for three cycles before the radiotherapy, and then receive radical radiotherapy(Intensive modulate radiotherapy,IMRT)and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy.
  Interventions: Drug: Paclitaxel liposome; Drug: Cisplatin; Drug: 5-fu; Radiation: Radical radiotherapy

INTERVENTIONS:
Drug: Paclitaxel liposome — Patients receive paclitaxel liposome(135mg/m2 on day 1),cisplatin (75mg/m2 Separate injection on day 1 to 3) and 5-fluorouracil (3750mg/m2 CIV 120h ) every three weeks for three cycl es before the radiotherapy.
  Patients receive radical radiotherapy and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy.
  Radical radiotherapy:Intensive modulate radiotherapy (IMRT),total dose for nasopharynx and nodule of neck:60Gy/30F,2.0Gy/daily.
  Other Names: Paclitaxel liposome,cisplatin,fluorouracil(TPF) chemotherapy
Drug: Cisplatin — Cisplatin (75mg/m2 Separate injection on day 1 to 3) with Paclitaxel liposome and 5-fu every three weeks for three cycles before the radiotherapy.Cisplatin(100mg/m2) every three weeks for three cycles during radiotherapy.
  Other Names: TPF induction chemotherapy; Concurrent cisplatin
Drug: 5-fu — Fluorouracil (3750mg/m2 CIV 120h)with Paclitaxel liposomeand cisplatin every three weeks for three cycles before the radiotherapy.
  Other Names: TPF induction chemotherapy
Radiation: Radical radiotherapy — Intensive modulate radiotherapy (IMRT) will be implement,total dose for nasopharynx and nodule of neck:60Gy(Gray)/30F(Fraction),2.0Gy/daily,5 days/week.
  Other Names: Concurrent radiotherapy

SUMMARY:
1. To see the effect if a combination of induction chemotherapy followed by chemoradiotherapy works in treating children with advanced nasopharyngeal carcinoma(NPC).

DETAILED DESCRIPTION:
This phase II trial is studying how well radiation therapy and chemotherapy work in treating young patients with newly diagnosed nasopharyngeal cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin and fluorouracil and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type).
* Original clinical staged as T4N0-3 M0 or any T、N3M0（according to the American Joint Committee on Cancer(AJCC) 7th edition）
* No evidence of distant metastasis (M0).
* Age ≤ 18 years old.
* Satisfactory performance status: Karnofsky scale (KPS) > 70.
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: creatinine clearance ≥60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age >18 years.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation.
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | After the completion of the chemoradiotherapy treatment (up to 9 weeks)
  CR assessed by independent reviewers, according to the Modified Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the chemoradiotherapy treatment. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) only

SECONDARY OUTCOMES:
Overall survival(OS) | 3-year
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Progress-free survival(PFS) | 3-year
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up
Locoregional failure-free survival(LRFS) | 3-year
  The LRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit
Distant metastasis-free survival(DMFS) | 3-year
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit
Short-term toxic effects assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0) | 3 months
  The shortterm toxic effects were assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0)
Long-term toxicities | Through study completion, an average of half year
  QoL was assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30)
Long-term toxicities | Through study completion, an average of half year
  EORTC quality of life questionnaire(QLQ) Head and Neck
Growth | Through study completion, an average of half year
  Patients will be monitored for height(in metre)
Growth | Through study completion, an average of half year
  Patients will be monitored for weight(in kilogram)
Growth | Through study completion, an average of half year
  Patients will be monitored for BMI(in kg/m^2)
Sex Development | Through study completion, an average of half year
  Sex hormone(estrogen,testosterone) levels(in nmol/L)
Sex Development | Through study completion, an average of half year
  Secondary sex characteristic survey
Intelligence Development | Through study completion, an average of half year
  Intelligence quotient by Stanford-Binet test

CONTACTS AND LOCATIONS:
Overall Officials: HaiQiang Mai, MD,PhD, Principal Investigator — Cancer center
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daoud J, Ghorbal L, Siala W, Elloumi F, Ghorbel A, Frikha M. [Is there any difference in therapeutic results of nasopharyngeal carcinoma between adults and children?]. Cancer Radiother. 2013 Dec;17(8):763-7. doi: 10.1016/j.canrad.2013.06.046. Epub 2013 Nov 20. French. PMID 24269016
- [Background] Yan Z, Xia L, Huang Y, Chen P, Jiang L, Zhang B. Nasopharyngeal carcinoma in children and adolescents in an endemic area: a report of 185 cases. Int J Pediatr Otorhinolaryngol. 2013 Sep;77(9):1454-60. doi: 10.1016/j.ijporl.2013.06.005. Epub 2013 Jul 3. PMID 23830224
- [Background] Liao WW, Tang SQ, Liu Y, Feng C. [Treatment of nasopharyngeal carcinoma in children]. Zhongguo Dang Dai Er Ke Za Zhi. 2013 Apr;15(4):273-6. Chinese. PMID 23607949
- [Background] Hu S, Xu X, Xu J, Xu Q, Liu S. Prognostic factors and long-term outcomes of nasopharyngeal carcinoma in children and adolescents. Pediatr Blood Cancer. 2013 Jul;60(7):1122-7. doi: 10.1002/pbc.24458. Epub 2013 Jan 9. PMID 23303571
- [Background] Cheuk DK, Billups CA, Martin MG, Roland CR, Ribeiro RC, Krasin MJ, Rodriguez-Galindo C. Prognostic factors and long-term outcomes of childhood nasopharyngeal carcinoma. Cancer. 2011 Jan 1;117(1):197-206. doi: 10.1002/cncr.25376. Epub 2010 Aug 24. PMID 20737561
- [Background] Buehrlen M, Zwaan CM, Granzen B, Lassay L, Deutz P, Vorwerk P, Staatz G, Gademann G, Christiansen H, Oldenburger F, Tamm M, Mertens R. Multimodal treatment, including interferon beta, of nasopharyngeal carcinoma in children and young adults: preliminary results from the prospective, multicenter study NPC-2003-GPOH/DCOG. Cancer. 2012 Oct 1;118(19):4892-900. doi: 10.1002/cncr.27395. Epub 2012 Feb 22. PMID 22359313
- [Background] Shen C, Gao Y, Xu T, Wang X, Ying H, Hu C. Carcinoma of the nasopharynx in young patients: a single institution experience. Clin Oncol (R Coll Radiol). 2009 Oct;21(8):617-22. doi: 10.1016/j.clon.2009.07.005. Epub 2009 Aug 5. PMID 19660923
- [Background] Varan A, Ozyar E, Corapcioglu F, Koksal Y, Aydin B, Yazici N, Akyuz C, Buyukpamukcu M. Pediatric and young adult nasopharyngeal carcinoma patients treated with preradiation Cisplatin and docetaxel chemotherapy. Int J Radiat Oncol Biol Phys. 2009 Mar 15;73(4):1116-20. doi: 10.1016/j.ijrobp.2008.05.028. Epub 2008 Sep 9. PMID 18786778
- [Background] Laskar S, Bahl G, Muckaden M, Pai SK, Gupta T, Banavali S, Arora B, Sharma D, Kurkure PA, Ramadwar M, Viswanathan S, Rangarajan V, Qureshi S, Deshpande DD, Shrivastava SK, Dinshaw KA. Nasopharyngeal carcinoma in children: comparison of conventional and intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):728-36. doi: 10.1016/j.ijrobp.2008.01.032. Epub 2008 Apr 18. PMID 18374512
- [Background] Selek U, Ozyar E, Ozyigit G, Varan A, Buyukpamukcu M, Atahan IL. Treatment results of 59 young patients with nasopharyngeal carcinoma. Int J Pediatr Otorhinolaryngol. 2005 Feb;69(2):201-7. doi: 10.1016/j.ijporl.2004.09.001. PMID 15656953
- [Background] Orbach D, Brisse H, Helfre S, Klijanienko J, Bours D, Mosseri V, Rodriguez J. Radiation and chemotherapy combination for nasopharyngeal carcinoma in children: Radiotherapy dose adaptation after chemotherapy response to minimize late effects. Pediatr Blood Cancer. 2008 Apr;50(4):849-53. doi: 10.1002/pbc.21372. PMID 17973328
- [Background] Ahern V, Jenkin D, Banerjee D, Greenberg M, Payne D. Nasopharyngeal carcinoma in the young. Clin Oncol (R Coll Radiol). 1994;6(1):24-30. doi: 10.1016/s0936-6555(05)80364-4. PMID 8172830
- See also: cisplatin — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: amifostine — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: paclitaxel — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: fluorouracil — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: nasopharyngeal carcinoma — http://www.nlm.nih.gov/medlineplus/
- See also: young patients — http://www.nlm.nih.gov/medlineplus/